CLINICAL TRIAL: NCT06987526
Title: Renewed Recovery: a Pilot Test of a Web-Based Mindfulness-Based Relapse Prevention Continuing Care Intervention for Individuals With Alcohol Use Disorder
Brief Title: Renewed Recovery: a Pilot Test of a Web-Based Mindfulness-Based Relapse Prevention Continuing Care Intervention for Alcohol Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PROJECT00011445
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Use Disorder (AUD)
Keywords: alcohol use disorder; recovery; continuing care; web-based; mindfulness-based relapse prevention; addiction
MeSH Terms: conditions — Alcoholism; Behavior, Addictive

STUDY DESIGN:
Intervention Model Description: This study uses a single-group, pre-post design to pilot test the feasibility, acceptability, and preliminary effects of a web-based Mindfulness-Based Relapse Prevention (MBRP) continuing care intervention ("Renewed Recovery") for individuals with alcohol use disorder (AUD) exiting standard outpatient treatment. Thirty participants will be enrolled and complete an 8-week self-guided web-based program. Assessments will be conducted at baseline, post-intervention, and 3-month follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Renewed Recovery Pilot Test (Experimental): Participants will complete an 8-week web-based Mindfulness-Based Relapse Prevention program delivered asynchronously. Each weekly module includes educational content, mindfulness exercises, and videos. In weeks 3 and 6, participants will also attend a live Zoom session led by the study's Co-Investigator for group meditation practice. Quantitative questionnaires will be delivered at program entrance, program completion, and 3 months post-program completion. A focus group will also be held at program completion.
  Prior to implementation, the intervention will be refined based on feedback from a usability test with individuals who have lived experience. The intervention content will be informed by a community needs assessment of treatment providers and individuals with AUD.
  Interventions: Behavioral: Mindfulness-Based Relapse Prevention

INTERVENTIONS:
Behavioral: Mindfulness-Based Relapse Prevention — Renewed Recovery is a web-based Mindfulness-Based Relapse Prevention (MBRP) continuing care intervention adapted from the original MBRP curriculum by Bowen et al. It consists of 8 weekly modules designed to teach mindfulness and relapse prevention strategies for individuals with alcohol use disorder. The intervention includes educational content, guided meditations, and practical exercises. Modules are delivered asynchronously online, supplemented by two live Zoom sessions for group meditation practice. The purpose of the curriculum is to teach mindfulness and relapse prevention techniques to the participants with the aim of reducing the risk for relapse. The module titles are as follows: (1) Automatic Pilot and Relapse, (2) Awareness of Triggers and Craving, (3) Mindfulness in Daily Life, (4) Mindfulness in High Risk Situations, (5) Acceptance and Skillful Action, (6) Seeing Thoughts as Thoughts, (7) Self-Care and Lifestyle Balance, and (8) Social Support and Continuing Practice.
  Other Names: MBRP

SUMMARY:
This study aims to design, implement, and evaluate a pilot test of a web-based Mindfulness-Based Relapse Prevention (MBRP) continuing care intervention to support individuals with alcohol use disorder (AUD) exiting standard outpatient treatment. Guided by the Centre for eHealth and Wellbeing Research (CeHRes) roadmap, the project follows a structured framework for digital intervention development: (1) contextual inquiry, (2) value specification, (3) design, (4) operationalization, and (5) summative evaluation. Contextual inquiry is defined as gathering information from the intended users and the environment in which the technology will be implemented. The next step, value specification, is defined as the quantification of the values of the key stakeholders, where the user requirements for the technology and the most favorable solutions emerge. This process elaborates on what was discovered in the contextual inquiry step and an analytical hierarchy is conducted to assign quantifiable values to the stakeholders' priorities for the intervention. Design is the step defined as the process of building prototypes of the technology that fit with the values and requirements of the stakeholders, and then testing the prototype in realistic situations. Operationalization is the implementation of the intervention. The final step, summative evaluation, is the assessment of the intervention's impact.

The research team plans to conduct a needs assessment (Aim 1a), develop (Aim 1b), implement (Aim 2a), and evaluate (Aim 2b) a pilot test of a web-based MBRP continuing care intervention, named "Renewed Recovery", targeting individuals exiting standard outpatient treatment for alcohol.

Aim 1: Design a web-based mindfulness continuing care intervention.

Aim 1a: Conduct a community needs assessment. To understand the need for such an intervention, semi-structured qualitative interviews with program administrators (n=3) from partnering substance use treatment facilities will be conducted (contextual inquiry). To better understand the recovery journey after exiting standard outpatient treatment, semi-structured interviews with individuals (n~10) who have been in treatment more than once will be conducted (contextual inquiry). After interviewing the 2 stakeholder groups, a meeting will be held to determine their list of priorities for this project (value specification).

Aim 1b: Develop the intervention website (design). The website for the intervention will be created by creating multiple wireframe iterations and presenting them to the stakeholders to determine the best formatting. The curriculum on the site will be modeled after the original MBRP curriculum. After coming to a consensus on the best version of the website, a usability test will be conducted of a newly created prototype with the same 10 individuals who identified as having been in treatment more than once. A quantitative survey will be employed and a focus groups will be held to assess the usability, equitability, enjoyability, and usefulness of the website.

Aim 2: Implement and evaluate the pilot test at partnering treatment facilities.

Aim 2a: Implement the pilot test of the web-based MBRP continuing care intervention (operationalization). After altering the intervention based on the usability test, the program will begin to be implemented. 30 people (3 groups of 10) will. Be recruited to participate in the intervention that will be 8 weeks in length (1 module per week, for a total of 8 modules), composed of a self-guided curriculum of text and videos, as well as two zoom sessions to practice meditating as a group.

Aim 2b: Evaluate the pilot test to determine process and behavior outcomes (summative evaluation). To measure process outcomes, surveys will be employed asking about the usability, equitability, enjoyability, and usefulness of the website as well as their overall satisfaction with the intervention. Recruitment and retention rates will be another identifier of process outcomes. To measure behavior outcomes, participants will be given a multitude of measures at baseline to measure relapse, anxiety, depression, self-efficacy, coping mechanisms, social support, acceptance, mindfulness, and reactivity to triggers. Analysis of these measures will be done via multilevel modeling. These measures will also be given at the completion of the program and at 3 months after completion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Currently leaving standard outpatient treatment within 1 week of the scheduled intervention start date, or has completed standard outpatient treatment within the past month
* Has access to the internet
* Scored 8 or above on the Alcohol Use Disorders Identification Test (AUDIT), or self-identifies as having been in treatment for alcohol use

Exclusion Criteria:

* Currently experiencing psychosis
* Currently experiencing dementia
* Does not have access to the internet
* Has not recently completed or left standard outpatient treatment within the specified timeline
* Does not meet criteria for alcohol use disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2026-03-22 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Alcohol consumption (Timeline Followback) | Baseline (program entry), 8 weeks (program completion), and 3-month follow-up
  Alcohol consumption will be assessed using the Timeline Followback (TLFB) method, a validated self-report instrument used to collect retrospective estimates of daily drinking.

SECONDARY OUTCOMES:
Substance Use (Timeline Followback) | Baseline (program entry), 8 weeks (program completion), and 3-month follow-up
  Substance use will be assessed using the Timeline Followback (TLFB), a validated self-report instrument used to collect retrospective estimates of daily drinking.
Depression (Short Form 6a PROMIS) | Baseline (program entry), 8 weeks (program completion), and 3-month follow-up
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Depression (Short form 6a) item bank assesses self-reported negative mood, views of self, and social cognition, as well as decreased positive affect and engagement. Higher scores indicate higher levels of depression. Minimum score = 38.4, maximum score = 80.3.
Anxiety (Short Form 8a PROMIS) | Baseline (program entry), 8 weeks (program completion), and 3-month follow-up
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety (Short Form 8a) item bank assesses self-reported fear, anxious misery, hyperarousal, and somatic symptoms related to arousal. Higher scores indicate higher levels of anxiety. Minimum score = 37.1, maximum score = 83.1.
Coping Behavior (Coping Strategies Inventory- Short Form) | Baseline (program entry), 8 weeks (program completion), and 3-month follow-up
  The Coping Strategies Inventory- Short Form (CSI-SF) is a self-reported instrument that assesses the prevalence of problem-focused and emotion-focused coping mechanisms. The measurement is broken down into 4 sub-scales: problem-focused engagement, problem-focused disengagement, emotion-focused engagement, and emotion-focused disengagement. Each sub-scale has a possible score range from 5 to 20. Higher scores on a sub-scale indicate greater use of that specific coping strategy by the participant.
Alcohol Cravings (Penn Alcohol Craving Scale) | Baseline (program entry), 8 weeks (program completion), and 3-month follow-up
  The Penn Alcohol Craving Scale (PACS) is a self-reported instrument that measures an individual's craving to drink alcohol. Scores range from 0 to 30. Higher scores indicate greater overall severity of alcohol craving.
Mindfulness (5 Facet Mindfulness Questionnaire) | Baseline (program entry), 8 weeks (program completion), and 3-month follow-up
  The 5 Facet Mindfulness Questionnaire (FFMQ) is a self-rated measurement on the five aspects of mindfulness namely: observation, description, aware actions, non-judgmental inner experience, and non-reactivity. Each facet is scored separately, with higher scores indicating greater levels of that particular mindfulness trait. Sub-scale scores can be analyzed individually or combined to reflect overall mindfulness, with higher total scores indicating greater overall mindfulness. For all facets except for non-reactivity, the score ranges from 8-40. For non-reactivity, the score ranges from 7-35.
Acceptance (Acceptance and Action Questionnaire II) | Baseline (program entry), 8 weeks (program completion), and 3-month follow-up
  The Acceptance and Action Questionnaire II (AAQII) measures psychological flexibility, defined as the ability to fully contact the present moment including all negative private events (which is thoughts, feelings, and physiological sensations) it contains, without needless defenses and depending on the situation engaging or changing behaviors in line with goals and values. Scores range from 7 to 49. Higher scores indicate less flexibility and acceptance, while lower total scores mean more flexibility.
Recovery Related Self-Efficacy (Alcohol Abstinence Self-Efficacy Scale) | Baseline (program entry), 8 weeks (program completion), and 3-month follow-up
  The Alcohol Abstinence Self-Efficacy Scale (AASE) is a self-reported instrument that assesses an individual's confidence in their ability to abstain from alcohol across a variety of high-risk situations. The scale consists of 20 items divided into four sub-scales representing different types of high-risk contexts: negative affect, social pressure, physical and other concerns, and withdrawal and urges. Higher scores on each sub-scale and the total score indicate greater self-efficacy in resisting the urge to drink alcohol in corresponding situations. The total score ranges from 20 to 100, while each sub-scale ranges from 5 to 25.
Triggers (Transaddiction Craving Triggers Questionnaire) | Baseline (program entry), 8 weeks (program completion), and 3-month follow-up
  The Transaddiction Craving Triggers Questionnaire (TCT) measures what kinds of things trigger the responder to have a craving for alcohol and/or substances. The questionnaire assesses various domains such as emotional states, environmental cues, social interactions, and physical sensations. There are three sub-scales: unpleasant affect (scores ranging from 14- 84), pleasant affect (scores ranging from 7-42), and cues and associated thoughts (scores ranging from 4-24). The total score ranges from 25-150. Higher total and sub-scale scores indicate a greater frequency of experiencing craving in response to specific types of triggers, reflecting higher craving vulnerability across those domains.
Social Support (Social Provisions Scale) | Baseline (program entry), 8 weeks (program completion), and 3-month follow-up
  The Social Provisions scale (SPS) is a measure of the provision of social support from current relationships. The scale is based on six provisions theorized to be critical to social support, making up the six sub-scales: guidance, reliable alliance, reassurance of worth, attachment, social integration, and opportunity for nurturance. The total score ranges from 24 to 96. Each sub-scale ranges from 4 to 16. Higher scores on the SPS indicate a greater perceived availability of social support across various domains. Higher sub-scale scores reflect stronger perceived support in that specific social domain.
Program Satisfaction (Client Satisfaction Questionnaire) | Program completion
  The Client Satisfaction Questionnaire (CSQ) is a self-rated instrument that asks participants to rate different aspects of the program to indicate their satisfaction with it. Participants rate various aspects of the program, such as quality of service, whether their needs were met, and their willingness to return or recommend the program. Scores range from 8 to 32. Higher total scores indicate greater overall satisfaction with the program.
Website Satisfaction (Systems Usability Scale) | Usability Test (formative/ Aim 1B) & Program completion (pilot test/Aim 2A)
  The System Usability Scale (SUS) is a 10-item self-reported questionnaire designed to assess the usability of a system, product, or digital platform. It measures overall user experience, including perceptions of ease of use, effectiveness, efficiency, and satisfaction. Scores range from 0 to 100. Higher scores indicate greater perceived usability of the system.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L Muilenburg, PhD, Principal Investigator — University of Georgia
Locations (2):
- United States (2):
  - Rescue Mission of Middle Georgia, Macon, Georgia
  - Project Adam, Winder, Georgia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data collected during the trial will be shared. This will include survey responses, program usage metrics, and outcome measures.
Time Frame: IPD will be available beginning 6 months after publication of the primary study results and will remain available for up to 5 years.
Access Criteria: Data will be made available to qualified researchers conducting ethically approved research. Requests will be reviewed by the study team for scientific merit and compliance with ethical standards.

REFERENCES:
- [Background] van Gemert-Pijnen JE, Nijland N, van Limburg M, Ossebaard HC, Kelders SM, Eysenbach G, Seydel ER. A holistic framework to improve the uptake and impact of eHealth technologies. J Med Internet Res. 2011 Dec 5;13(4):e111. doi: 10.2196/jmir.1672. PMID 22155738
- [Background] Bowen S, Chawla N, Collins SE, Witkiewitz K, Hsu S, Grow J, Clifasefi S, Garner M, Douglass A, Larimer ME, Marlatt A. Mindfulness-based relapse prevention for substance use disorders: a pilot efficacy trial. Subst Abus. 2009 Oct-Dec;30(4):295-305. doi: 10.1080/08897070903250084. PMID 19904665